CLINICAL TRIAL: NCT00597428
Title: A Multi-center, Randomized, Double-Blinded Study of the Efficacy and Safety of Lubiprostone in Patients With Opioid-induced Bowel Dysfunction (OBD)
Brief Title: Opioid-induced Bowel Dysfunction Pivotal Assessment of Lubiprostone
Acronym: OPAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sucampo Pharma Americas, LLC (Industry)
Collaborators: Sucampo Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mallinckrodt (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OBD0632
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Results first posted 2015-12-07 (Estimated); Last update posted 2019-12-10 (Actual); Status verified 2015-11

CONDITIONS: Opioid-Induced Bowel Dysfunction
MeSH Terms: conditions — Opioid-Induced Constipation | interventions — Lubiprostone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): 0 mcg capsules twice daily (BID)
  Interventions: Drug: Placebo
- Lubiprostone (Experimental): 24 mcg capsules twice daily (BID)
  Interventions: Drug: Lubiprostone

INTERVENTIONS:
Drug: Lubiprostone — 24 mcg capsules twice daily (BID)
  Other Names: Amitiza®
  Arms: Lubiprostone
Drug: Placebo — 0 mcg capsules twice daily (BID)
  Other Names: No other names
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to evaluate the efficacy and safety of lubiprostone administration in patients with opioid-induced bowel dysfunction (OBD).

ELIGIBILITY:
Inclusion Criteria:

* Consistent treatment for chronic, non-cancer-related pain with any full agonist opioid for at least 30 days prior to screening.
* Diagnosis of opioid-induced bowel dysfunction as confirmed during the screening period.
* If patient has a history of chronic constipation, condition must have been exacerbated by initiation of opioid treatment.
* Use of prescribed or over-the-counter (OTC) medication that affects gastrointestinal motility (other than opioid therapy) must be discontinued during the study.
* If treated for clinical depression with selective serotonin reuptake inhibitors (SSRIs), serotonin-norepinephrine reuptake inhibitors (SNRIs), or monoamine oxidase (MAO) inhibitors, treatment must have been at a stable dose for at least 30 days prior to screening.
* Use of laxative and stool softeners (with the exception of approved rescue medications) must be discontinued while on study.

Exclusion Criteria:

* Opioid dose adjustment (+/- 30%), and/or change in opioid agent or route of administration within 30 days of screening.
* Non-ambulatory patients, or those who are unable to eat/drink, take oral medications, or to hold down oral medications due to vomiting.
* Treatment with opioid therapy for cancer-related pain, abdominal pain, scleroderma, and/or for the management of drug addiction.
* Patient has been treated for cancer in the past 5 years (with the exception of localized basal cell, squamous cell skin cancer, or in situ cancer that has been resected).
* Gastrointestinal or abdominal surgical procedures within 90 days prior to screening.
* Female patients of childbearing potential who are unable/unwilling to use protocol-specified method(s) of birth control and/or are pregnant, nursing, or plan to become pregnant or nurse during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 437 (Actual)
Dates: Start 2007-08; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Egilius L.H. Spierings, M.D., Ph.D., Principal Investigator — MedVadis Research Corporation
Locations (114):
- United States (109):
  - Tuscaloosa VA Medical Center, Tuscaloosa, Alabama
  - Carl T Hayden VA Medical Center, Phoenix, Arizona
  - Redpoint Research, Phoenix, Arizona
  - HOPE Research Institute, LLC, Phoenix, Arizona
  - Clinical Research Advantage, Inc. / East Valley Family Physicians, PLC, Tempe, Arizona
  - Premiere Pharamaceutical Research, LLC, Tempe, Arizona
  - Harmony Clinical Research, Inc., Tucson, Arizona
  - Martin Bowen Hefley Knee, Little Rock, Arkansas
  - Advanced Pain Institute, Arcadia, California
  - Pain Institute of CA, Bakersfield, California
  - Catalina Research Institute, LLC, Chino, California
  - California Pain Center, Huntington Beach, California
  - Shreenath Clinical Service, Laguna Hills, California
  - Loma Linda University Physicians Medical Group, Loma Linda, California
  - VA Long Beach Healthcare System, Long Beach, California
  - Rider Research Group, San Francisco, California
  - Clinicos, LLC, Colorado Springs, Colorado
  - Rocky Mountain Gastroenterology Associates, Lakewood, Colorado
  - Arapahoe Gastroenterology, PC, Littleton, Colorado
  - Metro Clinical Research, LLC, Littleton, Colorado
  - Clinical Trial Management of Boca Raton, Inc., Boca Raton, Florida
  - Florida Institute of Medical Research, Jacksonville, Florida
  - Drug Study Institute, Jupiter, Florida
  - Gastroenterology Group of Naples, Naples, Florida
  - Kenneth W. Ponder, MD PA, Niceville, Florida
  - North Miami Research, Inc., North Miami, Florida
  - Renstar Inc., Ocala, Florida
  - Peninsula Research, Inc, Ormond Beach, Florida
  - DMI Research, Inc., Pinellas Park, Florida
  - Sunrise Medical Research, Inc., Plantation, Florida
  - Accord Clinical Research, LLC, Port Orange, Florida
  - Lovelace Scientific Resources, Inc., Sarasota, Florida
  - Meridien Research, St. Petersburg, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Advanced Pain Management, Augusta, Georgia
  - Global Research Partners & Consultants, Incs., Calhoun, Georgia
  - Q Clinical Research, Decatur, Georgia
  - Apex Medical Research, AMR, Inc., Chicago, Illinois
  - Claude Mandel Medical Center, Chicago, Illinois
  - Advanced Pain Care Clinic, Evansville, Indiana
  - MediSphere Medical Research Center, Evansville, Indiana
  - Davis Clinic, PC, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Louisville, Louisville, Kentucky
  - Gulf Coast Research, LLC, Lafayette, Louisiana
  - Delta Research Partners, LLC, Monroe, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Rehabilitation Team West, PA, Baltimore, Maryland
  - Columbia Medical Practice/ RxTrials, Inc., Columbia, Maryland
  - Washington County Hospital Association - The Center for Clinical Research, Hagerstown, Maryland
  - Beth Israel Deaconess Medical Center, Harvard Medical School, Boston, Massachusetts
  - MedVadis Research Corporation, Wellesley Hills, Massachusetts
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Professional Clinical Research, Inc., Interlochen, Michigan
  - PCM Medical Services, Lansing, Michigan
  - Women's Health Care Specialists, PC, Paw Paw, Michigan
  - Medical Research Associates, Traverse City, Michigan
  - Center for Digestive Health, Troy, Michigan
  - MAPS Applied Research Center, Edina, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Precise Research, Inc., Flowood, Mississippi
  - Medex Healthcare Research, St Louis, Missouri
  - Montana Neuroscience Institute Foundation / Montana Spine and Pain Center, Missoula, Montana
  - Creighton University Medical Center, Omaha, Nebraska
  - Advanced Biomedical Research of America, Las Vegas, Nevada
  - Lovelace Scientific Resources, Inc., Las Vegas, Nevada
  - Gastroenterology Research Associates, Cedar Knolls, New Jersey
  - Central Jersey Medical Research Center, Elizabeth, New Jersey
  - Holy Name Hospital, Institute for Clinical Research, Teaneck, New Jersey
  - Advanced Pain Consultants, Voorhees Township, New Jersey
  - Medex Healthcare Research, Inc., New York, New York
  - New York University Pain Management Center, New York, New York
  - Research Across America, New York, New York
  - North American Partners, Valley Stream, New York
  - Upstate Clinical Research Associates, Williamsville, New York
  - Randolph Medical Associates, Asheboro, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Carolina Research, Greenville, North Carolina
  - Carolina Digestive Health Associates, Harrisburg, North Carolina
  - Peters Medical Research, LLC, High Point, North Carolina
  - Triangle Medical Research, Lexington, North Carolina
  - Southern Gastroenterology Associates, New Bern, North Carolina
  - Valley Medical Primary Care, Centerville, Ohio
  - Glenway Family Medicine, Cincinnati, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Urgent Care Specialists, Dayton, Ohio
  - RAS Health Ltd., Marion, Ohio
  - University of Toledo - Health Science Campus, Toledo, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Paradigm Research Professionals, LLP, Oklahoma City, Oklahoma
  - Memorial Clinical Research, Oklahoma City, Oklahoma
  - Medford Medical Clinic, LLP, Medford, Oregon
  - Lehigh Valley Hospital - Neurosciences and Pain Research, Allentown, Pennsylvania
  - Einstein Pain Institute, Philadelphia, Pennsylvania
  - Jeffry A. Lindenbaum DO, PC, Yardley, Pennsylvania
  - Baptist Medical Tower Suite 740, Knoxville, Tennessee
  - Integrity Clinical Research, LLC, Milan, Tennessee
  - Texas Familicare Clinical Research, Hurst, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - Bexar Clinical Trials, LLC, Richardson, Texas
  - Advance Research Institute, Ogden, Utah
  - Highland Clinical Research, Salt Lake City, Utah
  - University of Utah, Salt Lake City, Utah
  - New River Valley Research Institute, Christiansburg, Virginia
  - Hampton Roads Institute for Performance and Sports Medicine (HIPS), Portsmouth, Virginia
  - McGuire Research Institute, Richmond, Virginia
  - Northwest Gastroenterology Associates, Bellevue, Washington
  - Daniel R. Coulston, Spokane, Washington
- Canada (5):
  - Hermitage Medicentre, Edmonton, Alberta
  - Health Sciences Centre, Winnipeg, Manitoba
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Pharmaceutical Integrated Research Company, London, Ontario
  - DHC Research, Richmond Hill, Ontario

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 06 August 2007 through 06 March 2009 Recruitment sites: 84 U.S. investigative sites and 4 Canadian investigative sites
Pre-assignment Details: Safety evaluable population (listed below under 'Started') includes all subjects who randomized and dosed. NOTE: these numbers are based on 1 miss randomized subjects - randomized to Lubiprostone and received Placebo. ITT population includes only those subjects who dosed and provided at least one post-treatment efficacy assessment.
Groups:
- Placebo: Placebo : 0 mcg capsules twice daily (BID) for 12 weeks
- Lubiprostone: Lubiprostone : 24 mcg capsules twice daily (BID) for 12 weeks
Period: Overall Study
Arm/Group | Placebo | Lubiprostone
Started | 214 | 223
Completed | 153 | 152
Not Completed | 61 | 71

BASELINE CHARACTERISTICS:
Population: Baseline analysis based on ITT population, which included 212 placebo-treated subjects and 223 lubiprostone-treated subjects.
Groups:
- Placebo: Placebo : 0 mcg capsules twice daily (BID)
- Lubiprostone: Lubiprostone : 24 mcg capsules twice daily (BID)
- Total: Total of all reporting groups
Arm/Group | Placebo | Lubiprostone | Total
Number analyzed (Participants) | 212 | 223 | 435
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (10.44) | 48.9 (9.85) | 49.4 (10.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126 | 140 | 266
  Male | 86 | 83 | 169
Region of Enrollment [Number; unit: participants]
  United States | 207 | 219 | 426
  Canada | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Weekly Spontaneous Bowel Movement (SBM) Frequency in Subjects Without Dose Reduction Prior to Week 8
Time Frame: Baseline and Week 8
Measure: Mean (Standard Deviation); unit: Spontaneous Bowel Movements/Week
Arm/Group | Placebo | Lubiprostone
Number analyzed (Participants) | 212 | 223
Spontaneous Bowel Movements/Week | 2.4 (3.20) | 2.6 (3.26)

2. Secondary Outcome: Change From Baseline in Mean Weekly SBM Frequency
Description: For overall assessment of change, average weekly rating was calculated from data collected from Week 1 through Week 12.
Time Frame: Baseline, Week 12, and Weeks 1-12
Measure: Mean (Standard Deviation); unit: Spontaneous Bowel Movements/Week
Arm/Group | Placebo | Lubiprostone
Number analyzed (Participants) | 209 | 217
Spontaneous Bowel Movements/Week
  Week 12 | 2.6 (3.57) | 2.5 (3.64)
  Overall | 2.3 (2.57) | 2.6 (2.73)

3. Secondary Outcome: First Post-dose SBM
Description: The number of participants that experienced first post-dose SBM 24 and 48 hour of dose initiation.
Time Frame: 24 and 48 hours post-dose
Measure: Number; unit: participants
Arm/Group | Placebo | Lubiprostone
Number analyzed (Participants) | 212 | 223
participants
  24 hours | 64 | 74
  48 hours | 118 | 136

4. Secondary Outcome: Responder Rate
Description: Number of participants, who remained on treatment for at least 8 weeks, and reported response (>=3 SBMs) for at least 50% of weeks on study.
Time Frame: Up to 12 weeks
Measure: Number; unit: participants
Arm/Group | Placebo | Lubiprostone
Number analyzed (Participants) | 212 | 223
participants | 100 | 108

5. Secondary Outcome: Mean Changes From Baseline in Straining, Stool Consistency, Constipation Severity, Abdominal Bloating, Abdominal Discomfort, and Bowel Habit Regularity
Description: Ratings over 12-week treatment period were averaged and difference from baseline score calculated Straining scale: 0 = absent, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe Stool consistency scale: 0 = very loose, 1 = loose, 2 = normal, 3 = hard, 4 = very hard (little balls) Constipation severity scale: 0 = absent, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe Abdominal bloating scale: 0 = absent, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe Abdominal discomfort scale: 0 = absent, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe Bowel habit regularity scale: 7-point scale, where 1 = very regular and 7 = very irregular
Time Frame: Weeks 1-12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lubiprostone
Number analyzed (Participants) | 212 | 223
units on a scale
  Straining | -0.5 (0.89) | -0.8 (0.96)
  Stool consistency | -0.4 (0.81) | -0.6 (0.84)
  Constipation severity | -0.5 (0.72) | -0.6 (0.79)
  Abdominal bloating | -0.4 (0.64) | -0.5 (0.70)
  Abdominal discomfort | -0.4 (0.64) | -0.5 (0.69)
  Bowel habit regularity | -0.6 (1.57) | -0.8 (1.57)

6. Secondary Outcome: Treatment Effectiveness
Description: Treatment effectiveness scale: 0 = not at all effective, 1 = a little bit effective, 2 = moderately effective, 3 = quite a bit effective, 4 = extremely effective
Time Frame: Weeks 1-12
Population: Treatment effectiveness scores were collected at the end of each treatment week during the study; the number of participants analyzed reflects those subjects who provided at least one end-of-week assessment of treatment effectiveness. For the analysis, treatment effectiveness scores were averaged across the treatment period (Weeks 1-12).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lubiprostone
Number analyzed (Participants) | 201 | 213
units on a scale | 1.4 (1.04) | 1.5 (1.07)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (AEs): 13 weeks (from time of first dose to 7 days post-treatment)
Description: Number of participants at risk represents the Safety Evaluable population. Safety Evaluable population includes all subjects who randomzied and dosed. ITT population (in Participant Flow) includes only subjects who dosed and provided at least one post-treatment efficacy assessment.
Arm/Group | Placebo | Lubiprostone
Serious Adverse Events (participants affected / at risk) | 7/214 | 7/223
Other Adverse Events (participants affected / at risk) | 36/214 | 49/223
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=214) | Lubiprostone (N=223)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Faecaloma (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Multiple sclerosis relapse (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Tricuspid valve disease (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Chills (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=214) | Lubiprostone (N=223)
Nausea (Gastrointestinal disorders) | 19 | 33
Diarrhoea (Gastrointestinal disorders) | 9 | 18
Flatulence (Gastrointestinal disorders) | 9 | 13
Vomiting (Gastrointestinal disorders) | 7 | 12

LIMITATIONS AND CAVEATS:
Post-study, it was determined that lubiprostone efficacy was dose-dependently decreased with concomitant methadone use (30% higher morphine equivalent daily dose (MEDD) than parallel pivotal study NCT00595946).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days